CLINICAL TRIAL: NCT03890484
Title: Peer Groups and Broad Social Motives' Influence on College Student Drinking: A Multimethod Approach Using Alcohol Administration and Daily Diary
Brief Title: The College, Alcohol and Peers Study (CAPS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment due to COVID pandemic; termination of funding
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mary Larimer, Professor, School of Medicine, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006279; F31AA027471-01 (NIH)
Record Dates: First submitted 2018-12-20; First posted 2019-03-26 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Alcohol Drinking
Keywords: Alcohol use; Risk-taking; Anxiety; Motives; Multimethod
MeSH Terms: conditions — Alcohol Drinking; Risk-Taking; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions, which will run in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Peers (Experimental): Participants will drink with two new peers (i.e. strangers), who they did not know prior to the study and their Peer Type.
  Interventions: Behavioral: Peer Type - New Peer
- Close Friends (Experimental): Participants will recruit and drink with two of their close friends and their Peer Type
  Interventions: Behavioral: Peer Type - Close Friends

INTERVENTIONS:
Behavioral: Peer Type - New Peer — Participants drink with 2 unfamiliar confederate peers
  Arms: New Peers
Behavioral: Peer Type - Close Friends — Participants drink with 2 close friends
  Arms: Close Friends

SUMMARY:
The present study will evaluate college students (N=100) from 2- and 4-year colleges/universities between 21-24 years old to assess anxiety, affect, broad social motives (BSM) and peer group influences on drinking and other risk-taking behaviors. This study will employ two sound scientific methods for testing behavior during drinking events (i.e., lab alcohol administration and daily diary) and use novel strategies to compare results of these two methods in the same sample. Using an ad-lib drinking paradigm, students' risk-taking, as measured by the Balloon Analogue Risk Task (BART), will be assessed when alone and during one of two randomly assigned peer group conditions (close friends or new peers). Participants will be allowed to freely drink (within safety limits) with their peer group prior to completing the BART again. These same students will complete daily electronic diaries on four weekends (Thursday - Sunday; total 24 assessments) regarding BSM, motives to drink, peers in their social group, alcohol use and consequences, and if/how their social group changed (e.g., few close friends to large party with many new peers) during the drinking event. Competing hypotheses will be tested such that: 1) anxiety is expected to be a stronger predictor of drinking behavior and greater differences in risk-taking in the new peer condition than close friend condition or 2) BSM is expected to be a stronger predictor of drinking behavior and greater differences in risk-taking in the close friend condition than new peers condition. Results are expected to be replicated in the daily diary reports. Further, this multimethod approach will allow us to evaluate how behavior assessed in the lab predicts naturally occurring behaviors in an uncontrolled setting. For example, the investigators will assess whether greater increases in self-reported risk-taking from baseline to after entering peer groups in the bar lab setting will predict heavier drinking on nights when most drinking companions are close friends reported during daily diary.

DETAILED DESCRIPTION:
Participants (N=100) will be recruited through direct outreach to University of Washington (UW) students via the UW Registrar's directory list, as well as community flyers distributed at colleges in the local area, online advertisements, and word of mouth. Participants will complete screening measures online. Eligible participants will be stratified on sex, age, and past 30-day peak alcohol use and randomly assigned to one of two conditions: close friends (N=50), where participants will recruit two of their existing friends, or new peers (N=50), where participants will drink with two strangers. To ensure at least two eligible friends, those in the close friend group will be asked to provide email and phone numbers of five to seven close friends. Close friends will have to meet the same inclusion and exclusion criteria as target participants and will go through the same procedures as target participants during alcohol administration. For each pair of participants matched on the three strata (age, sex, alcohol use), strangers in the new peer group will be matched to the sex of the close friends of the other matched participant's group.

Participants will be asked not to travel to the bar together to ensure they are not exposed to their peer group before entry to the bar, and must get to the lab without operating any vehicle with wheels (e.g. car, bike). Upon arriving to the lab, all participants and peers will review and sign the consent form, and provide a baseline breath alcohol content (BrAC) reading. Female participants and friends will also be asked to take a urine pregnancy test. Participants and friends will complete baseline measures and the Balloon Analogue Risk Task (BART) individually prior to entry to the bar. Then they will be taught the procedures for the daily diary portion of the study (see below). Participants will join their close friends or new peers in the bar and be given 20 minutes to relax while the researcher prepares the materials. After entering groups but prior to receiving alcohol, participants and peers will complete pre-alcohol measures and the BART. They will then be allowed to order anything from the bar menu for the following hour. Participants and close friends will be allowed to drink freely within limits (BrAC = .12%), for safety. During ad-lib, estimated BAC levels based on age, sex, and weight will be calculated prior to each drink served to ensure the safety of consuming each drink without interrupting social interaction and making the participant's BAC more salient by taking BrAC readings regularly. Participants or close friends whose BAC may exceed .12% will only be served placebo beverages for the remainder of the hour. BrAC readings will be taken at the end of ad-lib, every 10 minutes until peak BrAC is reached and readings are descending, and every 30 minutes thereafter. After ad-lib, participants will complete post-alcohol measures and the BART, then provided entertainment until they reach a BAC below .03%. The full protocol will take approximately 2.5 hours. On average, alcohol metabolizes at a rate of .015% per hour, so a participant who reaches .12% will be in the lab on average 8.5 hours. Once sober, participants and friends will be taken home in a taxi or ride share service (e.g. Uber, Lyft). Close friends will not complete the following daily diary protocols.

Daily diary measures will start on the Thursday following each participant's alcohol administration appointment and be collected for potential drinking events on Thursday, Friday, and Saturday over the following four consecutive weeks. Each day, participants will be notified of surveys by text message at 4 pm and the following morning at 11am (Friday, Saturday, and Sunday) for a total of 24 assessments. Surveys will be available for 2 hours and reminders sent via text 30 minutes before closing. Afternoon assessments take approximately 5 minutes and measure BSM, motives to drink, motives to refrain from drinking, evening plans, and what type of peers they plan to spend the evening with (e.g. close friends, new peers, family, alone). For the daily diary, BSM items have been modified to select experiences which may vary daily (e.g. "making social plans got me excited and energized today) and drinking motives have been modified into a brief prospective measure consistent with modifications used in other studies15. At morning assessments, participants will retrospectively report amount of drinks and other substances consumed, time spent drinking, and consequences experienced while drinking or currently (morning after drinking). Participants will be asked how many times their social group changed during the event defined as the majority of their drinking companions being of a different peer type than before. For instance, a participant may be at a house party with primarily close friends, but someone invites several people the participant does not know well and they are now drinking with mostly new peers. For each peer group reported (up to five groups), participants will report the following characteristics of the group: size (i.e. number of people they had direct contact with), number of drinking companions of each peer type (e.g. close friends, new peers, family), gender composition of the group (same-sex vs. mixed-sex), time spent with and drinks consumed with each group. On non-drinking evenings, participants will report similar information regarding their social groups and other activities. This survey will take approximately 5-7 minutes.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled in college
* has consumed 3 or more alcoholic drinks in one sitting at least once in the past month
* drinking frequency of once a week

Exclusion Criteria:

* past-month alcohol
* past-month other substance dependence,
* past-month mood disorder
* past-month anxiety disorder
* past-moth suicidal ideation
* excessive alcohol use reaching a BAC greater than .30% in past month
* history of serious medical conditions
* regular use of prescription psychotropic or pain medication
* history of negative reactions to alcohol
* history of treatment for alcohol use disorder
* pregnancy
* nursing

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2022-07-03 (Actual); Study Completion 2022-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Larimer, PhD, Principal Investigator — University of Washington
Locations (1):
- The Center for the Study of Health and Risk Behaviors, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through University registrar's list emails, flyers posted around campus, and social media advertisements. Participants were recruited and enrolled between December 2019 and July 2022. Recruitment was paused from March 2020 to August 2021 due to the COVID-19 pandemic and again from August 2022 until early termination in June 2023 due to key personnel and funding changes. Study effective termination was July 2022.
Pre-assignment Details: Participants were completed informed consent and enrolled at the time of the alcohol administration session.
Period: Overall Study
Arm/Group | New Peers | Close Friends
Started | 5 | 8
Completed Alcohol Admin Session | 5 | 8
Completed | 4 | 7
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled completed Baseline
Groups:
- Total: Total of all reporting groups
Arm/Group | New Peers | Close Friends | Total
Number analyzed (Participants) | 5 | 8 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 8 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (0.89) | 21.5 (0.76) | 21.46 (0.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 7 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 8 | 13
Broad Social Motives for Friends [Mean (Standard Deviation); unit: units on a scale] — Measures reward responsiveness towards social interactions with friends. Measured by 21 items on a 5-point Likert scale ranging from 1 = Strongly disagree to 5 = strong agree. Mean scores were created from all items. Higher values are better.
  units on a scale | 4.06 (0.44) | 4.58 (0.32) | 4.38 (0.44)
Broad Social Motives for New Peers [Mean (Standard Deviation); unit: units on a scale] — Measures reward responsiveness toward social interactions with strangers and people just meeting for the first time. Measures by 20 items on a 5 point Likert scale ranging from 1 = strong disagree to 5 = strongly agree. Mean scores were created from all items. Higher values are better.
  units on a scale | 2.87 (0.23) | 3.94 (0.51) | 3.53 (0.68)
Negative Affect [Mean (Standard Deviation); unit: units on a scale] — The state version of the Positive and Negative Affect Scale (PANAS; Watson, Clark, & Tellegen, 1988) is a 20-item measure. All adjectives reflect positive (e.g., excited) or negative (e.g., hostile) feeling words. Response options are rated on a 5-point Likert scale from 0 = "Very slightly or not at all" to 4 = "Extremely". Mean scores were created from all items. Lower values are better.
  units on a scale | 1.4 (0.27) | 1.11 (0.14) | 1.22 (0.24)
Positive Affect [Mean (Standard Deviation); unit: units on a scale] — The state version of the Positive and Negative Affect Scale (PANAS; Watson, Clark, & Tellegen, 1988) is a 20-item measure. All adjectives reflect positive (e.g., excited) or negative (e.g., hostile) feeling words. Response options are rated on a 5-point Likert scale from 0 = "Very slightly or not at all" to 4 = "Extremely". Mean scores were created from all items. Higher values are better.
  units on a scale | 2.7 (0.68) | 3.16 (0.50) | 2.98 (0.60)
Prior 30 day Alcohol Consequences [Mean (Standard Deviation); unit: units on a scale] — The Young Adult Alcohol Problem Screening Test (YAAPST; Hurlbut & Sher, 1992) includes 27 items measuring frequency of experiencing negative alcohol consequences. Frequency options vary by item, please see Hurlbut & Sher, 1992 for full scoring instructions. A sum score was created as a consequence severity score. The scale can range from 0 to 134. Lower scores are better.
  units on a scale | 16.2 (6.72) | 20 (15.76) | 18.54 (12.79)
Prior 30 day Alcohol Use [Mean (Standard Deviation); unit: Number of standard drinks] — The Time-Line Follow Back (TLFB; Sobell & Sobell, 1992) is a semi-structured interview to collect details of drinking events over the past month. Average number of standard drinks was calculated for results.
  Number of standard drinks | 2.91 (0.93) | 3.04 (1.15) | 2.99 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Number of drinks consumed
Time Frame: During 1 hour ad-lib period, starting an average of 1 hour after Baseline.
Measure: Mean (Standard Deviation); unit: Number of drinks
Arm/Group | New Peers | Close Friends
Number analyzed (Participants) | 5 | 8
Number of drinks | 3.2 (0.45) | 3.63 (0.74)

2. Primary Outcome: Alcohol Use - Daily Diary
Description: Number of drinks consumed, self-reported the morning after drinking events
Time Frame: 4 weeks following ad-lib.
Measure: Mean (Standard Deviation); unit: Number of drinks
Arm/Group | New Peers | Close Friends
Number analyzed (Participants) | 4 | 7
Number of drinks | 3.8 (2.57) | 2.61 (1.7)

3. Primary Outcome: Alcohol Consequences
Description: Self-report of the Young Adult Alcohol Problems Screening Test (YAAPST). Count of number of consequences experienced. Range: 0-27. Higher scores represent more consequences experienced.
Time Frame: 4 weeks following ad-lib.
Measure: Mean (Standard Deviation); unit: Number of consequences
Arm/Group | New Peers | Close Friends
Number analyzed (Participants) | 4 | 7
Number of consequences | 0.40 (0.74) | 0.30 (0.56)

4. Primary Outcome: Risk-taking
Description: Scores on the Balloon Analogue Risk Task (BART). Scores are calculated by adding the number of pumps for unexploded balloons, with higher scores reflecting greater risk-taking. Range varies - explosions are at a random point between 1 and 128 pumps.
Time Frame: Change from baseline (alone) to 20 minutes following Peer Type intervention.
Measure: Mean (Standard Deviation); unit: Number of pumps
Arm/Group | New Peers | Close Friends
Number analyzed (Participants) | 5 | 8
Number of pumps | 8.02 (9.57) | 15.29 (19.83)

5. Primary Outcome: Risk-taking
Description: as for outcome 4
Time Frame: Change from baseline (alone) to immediately following ad-lib, an average of 2 hours after baseline.
Measure: Mean (Standard Deviation); unit: Number of pumps
Arm/Group | New Peers | Close Friends
Number analyzed (Participants) | 5 | 8
Number of pumps | 12.83 (10.77) | 28.27 (21.11)

ADVERSE EVENTS:
Time Frame: One month
Description: All-Cause Mortality was not monitored during the 4-week follow-up period because all assessments were self-reported. Mortality would have only been reported to study staff if the participant's next of kin choose to share that information.
  Serious adverse events monitored was consuming alcohol at potentially lethal doses of BAC > .30.
  Other non-serious adverse events monitored was becoming nauseous by self-report or exceeding a BrAC > .15 during alcohol administration procedures.
Arm/Group | New Peers | Close Friends
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 0/5 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03890484/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03890484/SAP_001.pdf